CLINICAL TRIAL: NCT02560701
Title: Impact of High Deductible Health Plans on Patients With Bipolar Disorder
Brief Title: High Deductible Health Plans and Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Depression and Bipolar Support Alliance (Unknown); NAMI: National Alliance on Mental Illness (Unknown)
Responsible Party: Sponsor
Other Study IDs: IHS-1408-20393
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2019-05

CONDITIONS: Bipolar Disorder
Keywords: high-deductible health plans; medication adherence
MeSH Terms: conditions — Bipolar Disorder; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Patient Interview — Investigators will conduct in-depth interviews with approximately 40 commercially insured individuals with bipolar disorder or their family caregivers to explore how they navigate deductibles, copayments, and other complex insurance features. Investigators will also determine the health care services that patients most value and assess how they prioritize difficult health care cost tradeoffs.

SUMMARY:
Using eleven years (2004-2014) of claims data from the largest US commercial health insurer, the investigators will assess the impact of switching into high-deductible health plans (HDHPs) on outcomes for patients with bipolar disorder. Patient subgroups will include patients with and without high medication cost-sharing and vulnerable populations (racial/ethnic minorities, poor, rural, major comorbidities). Interviews with patients and caregivers recruited through a major advocacy group will provide further insights into the policy issues with real-life experiences.

DETAILED DESCRIPTION:
Bipolar disorder is a severe mental illness affecting about 3% of the U.S. population that causes personal suffering, morbidity, and premature mortality. Continuous access to medications, close monitoring, and other psychiatric care are crucial for avoiding complications of bipolar disorder such as relapse, hospitalization, and suicide. To control rising costs, payers and employers are increasingly adopting high-deductible health plans (HDHPs) with very high out-of-pocket payments. Federally-defined Health Savings Account HDHPs require full cost-sharing for all non-preventive services, including medications and specialist visits; family deductibles for HSA-HDHPs range from $2,500 to $12,700. Enrollment in HDHPs quadrupled nationally between 2006 and 2013 to 38% of all workers. Analysts expect further explosive growth because of continued health care cost pressure on families and employers. Well-informed patients in HDHPs might reduce use of unnecessary services and more expensive treatment options. However, patients might also choose to forego needed care. There is very little evidence on how particularly vulnerable patients such as those with bipolar disorder or other chronic mental illnesses fare when forced to make complex choices about spending for care under HDHPs. Given their rapid escalation, there is an urgent need to understand how vulnerable patients change their patterns of care and medication adherence under HDHPs. We will compare patients with three types of insurance: traditional plans with low or no deductible; HDHPs in which chronic medications are paid fully out-of-pocket until the deductible is met; and HDHPs where medications are subject to the same co-pays as in traditional plans.

OBJECTIVES:

Using ten years of data from the largest U.S. commercial health insurer (~70 million members in all 50 states), we will assess the impact of HDHPs on key outcomes for patients with bipolar disorder experiencing employer-mandated shifts from traditional insurance to HDHPs. Our specific aims are to evaluate: (1) changes in medication adherence, and in intensity and quality of other health care; (2) changes in adverse events; and, (3) changes in patient out-of-pocket costs. We will compare how these outcomes differ for patients in HDHPs with and without medications subject to the deductible. We will assess effects in the overall population of patients with bipolar illness and in specific vulnerable subgroups, including racial/ethnic minorities, poorer patients, rural patients, and patients with other important comorbidities.

METHODS:

We will take advantage of an ongoing natural experiment whereby employers have shifted all their employees at once from traditional insurance to HDHPs. We will use the strongest quasi-experimental, longitudinal methods available to compare the experience of patients switched by their employers into HDHPs with contemporaneous patients whose employers remain in traditional plans. A major advantage of our approach is the inclusion of only employers whose employees had no choice of insurance plans, minimizing member-level selection bias.

From preliminary data queries, we estimate a study population of ~160,000 members with bipolar disorder from 2004-2013. Our data include detailed information about insurance type, diagnoses, health services and pharmacy utilization, out-of-pocket payments, individual-level patient characteristics like income, and neighborhood-level factors like racial density. The unprecedented large sample size will allow us to answer questions about how patients from particular vulnerable subgroups respond to HDHPs, including patients who are Black or Hispanic, have low incomes, reside in rural areas, and have major comorbidities.

PATIENT OUTCOMES:

Our Aim 1 measures of the quality of bipolar treatment will include indicators of patients' access to appropriate care: prevalence and intensity of use of effective medications (antipsychotics, anticonvulsants); medication adherence; and, guideline-recommended clinical monitoring (regular outpatient mental health visits). Adverse events in Aim 2 will include psychiatric hospitalizations, which are potentially avoidable and often viewed as an indicator of suboptimal outpatient care. In Aim 3, we will assess changes under HDHPs in the co-payment amounts faced by patients for specific medical services, such as prescription fills and clinician visits, and the total burden of patient out-of-pocket costs.

PATIENT AND STAKEHOLDER ENGAGEMENT:

Our longstanding engagement with the National Alliance on Mental Illness (NAMI, the preeminent patient advocacy organization addressing issues around bipolar disorder) has shaped our study aims and our focus on measurable outcomes of particular concern to patients. We will solicit regular input from a local patient and family advisory panel (assembled with NAMI's assistance) on the refinement of methods, interpretation of study findings, shaping of recommendations, and dissemination of results. As study consultant, NAMI Medical Director Dr. Ken Duckworth will guide meetings of the patient panel and contribute perspectives from the broader community of patients and clinicians dealing with bipolar illness. Dr. Greg Simon, Director of the US Mental Health Research Network, will provide national expertise on patient experiences with serious mental illness in health plans.

ANTICIPATED IMPACT:

Our research will provide empirical data comparing how patients with bipolar illness fare under three insurance designs with vastly different requirements for cost-sharing. At a time when HDHP enrollment is exploding, the experience of patients with serious mental illnesses is largely unexamined. Advocacy groups will be able to use our findings to lobby for more patient-responsive benefit designs; policymakers will have evidence to redesign insurance benefits to better address the needs of vulnerable patients (e.g., by exempting mood stabilizing agents from deductibles).

ELIGIBILITY:
Inclusion Criteria (for both study intervention/control groups):

[Intervention Cohort]:

* Traditional plan members with bipolar illness.
* Experience an employer-mandated switch to HSA-eligible HDHPs with full drug cost-sharing.

[Control Cohort]:

* Members with bipolar illness.
* Members whose employers offered only a traditional plan for the follow-up year.

Exclusion Criteria:

* Members age 65 years or older who could be eligible for Medicare benefits, including drug coverage through Medicare Part D.
* Members whose employer offered a choice of health plan.

Ages: 12 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Investigators will include health plan members aged 12 to 63 years at the beginning of the baseline period. Consistent with prior research,89-91 we will use medical claims data and a validated algorithm to identify members who had at least two ambulatory encounters or one hospital encounter with a diagnosis of bipolar disorder. Intervention cohorts will include traditional plan members with bipolar illness who experience an employer-mandated switch to HSA-eligible HDHPs with full drug cost-sharing or to HSA-ineligible HDHPs that subject medications only to copayments as in traditional health plans.
Sampling Method: Non-Probability Sample
Enrollment: 350823 (Actual)
Dates: Start 2015-09; Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Wharam, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute

IPD SHARING:
Plan to Share IPD: No
Per contract with our data vendor, we are unable to share individual participant data but will maintain records internally in accordance with funder guidelines.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified in claims data. Each was required to have one inpatient episode or two outpatient visits with a corresponding diagnosis of bipolar disorder. Patients with schizophrenia or schizoaffective disorder were excluded.
Pre-assignment Details: Study participants without either a) two years of continuous enrollment in a low-deductible health plan OR b) one year of enrollment in a low-deductible plan followed by a continuous year of enrollment in a high-deductible plan were excluded. This brought the sample size from 350,823 to 97,302.
Groups:
- High-Deductible Health Plan Group: Insurance plan members with one year in a low-deductible plan (less than or equal to $500 per year), followed by an employer mandated switch to a high-deductible plan (greater than or equal to $1,000 per year)
- Control Group: Insurance plan members with two consecutive years in employer-mandated low-deductible plans (less than or equal to $500 per year)
Period: Overall Study
Arm/Group | High-Deductible Health Plan Group | Control Group
Started | 8060 | 89242
Carve Out (Patients in employers who carved out mental health insurance coverage to a 3rd party vendor excluded) | 8060 | 88729
Restrict to Patients Between 12 and 64 | 7598 | 82367
Bipolar Diagnosis Time Constraints (Require most recent bipolar diagnosis to be between 5 years and 4 months prior to intervention date) | 3533 | 39427
Matched Cohort | 3517 | 37776
Completed | 3517 | 37776
Not Completed | 4543 | 51466

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Deductible Health Plan Group | Control Group | Total
Number analyzed (Participants) | 3517 | 37776 | 41293
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (13.7) | 38.3 (14.1) | 38.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 10 participants in control group were missing gender information
  Participants
    number analyzed (Participants) | 3517 | 37766 | 41283
    Female | 2130 | 23153 | 25283
    Male | 1387 | 14613 | 16000
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 126 | 1458 | 1584
  Not Hispanic or Latino | 3391 | 36318 | 39709
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 519 | 557
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 422 | 451
  White | 2599 | 25982 | 28581
  More than one race | 685 | 8701 | 9386
  Unknown or Not Reported | 166 | 2152 | 2318
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Midwest | 1203 | 11003 | 12206
  United States: Northeast | 253 | 4720 | 4973
  United States: South | 1616 | 16283 | 17899
  United States: West | 445 | 5770 | 6215
Substance Use Disorder Flag [Count of Participants; unit: Participants]
  Substance Use Disorder | 638 | 6283 | 6921
  No Evidence of Substance Use Disorder | 2879 | 31493 | 34372
Rural [Count of Participants; unit: Participants]
  Non-Urban | 258 | 2492 | 2750
  Urban | 3259 | 35284 | 38543

OUTCOME MEASURES:

1. Primary Outcome: Inpatient Hospitalizations Among Bipolar Patients
Description: Mean number of annual inpatient hospitalizations in the follow-up period among bipolar patients
Time Frame: Year 3
Measure: Mean (Standard Deviation); unit: hospitalizations per year
Arm/Group | High-Deductible Health Plan Group | Control Group
Number analyzed (Participants) | 3517 | 37776
hospitalizations per year | 0.17 (0.60) | 0.17 (0.57)

2. Primary Outcome: Emergency Department Visits Among Patients With Bipolar Disorder
Description: Mean number of annual emergency department visits in the follow-up period among bipolar patients
Time Frame: Year 3
Measure: Mean (Standard Deviation); unit: ED visits per year
Arm/Group | High-Deductible Health Plan Group | Control Group
Number analyzed (Participants) | 3517 | 37776
ED visits per year | 0.42 (1.26) | 0.38 (1.09)

3. Primary Outcome: Medication Adherence for Bipolar Disorder
Description: Mean number of annual bipolar medication fills in the follow-up period among bipolar patients
Time Frame: YEAR 2
Measure: Mean (Standard Deviation); unit: Medication fills per year
Arm/Group | High-Deductible Health Plan Group | Control Group
Number analyzed (Participants) | 3517 | 37776
Medication fills per year | 0.57 (3.15) | 1.42 (4.47)

4. Secondary Outcome: Access To Outpatient Services for Bipolar Disorder
Description: Mean number of annual outpatient mental health visits for bipolar patients, averaged across baseline and follow-up periods
Time Frame: YEAR 2
Measure: Mean (Standard Deviation); unit: visits per year
Arm/Group | High-Deductible Health Plan Group | Control Group
Number analyzed (Participants) | 3517 | 37776
visits per year | 5.54 (8.48) | 6.15 (9.54)

5. Other Pre Specified Outcome: Annual Patient Out-of-pocket Costs for Patients With Bipolar Disorder
Description: Annual patient out-of-pocket costs (paid deductible, coinsurance, and copayment amounts) for patients with Bipolar Disorder in the baseline period
Time Frame: YEAR 2, YEAR 3
Measure: Mean (Standard Deviation); unit: U.S. Dollars per year
Arm/Group | High-Deductible Health Plan Group | Control Group
Number analyzed (Participants) | 3517 | 37776
U.S. Dollars per year | 1674.61 (1576.04) | 1440.45 (1510.86)

6. Secondary Outcome: Medication Adherence for Bipolar Disorder - Psychotropic Medications
Description: Mean number of annual psychotropic medication fills in the follow-up period among bipolar patients
Time Frame: YEAR 2
Measure: Mean (Standard Deviation); unit: medication fills per year
Arm/Group | High-Deductible Health Plan Group | Control Group
Number analyzed (Participants) | 3517 | 37776
medication fills per year | 0.73 (3.73) | 2.57 (6.92)

ADVERSE EVENTS:
Time Frame: 3 years
Description: This study was conducted retrospectively using claims data. Adverse events are not applicable to this study design.
Arm/Group | High-Deductible Health Plan Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/3517 | 0/37776
Serious Adverse Events (participants affected / at risk) | 0/3517 | 0/37776
Other Adverse Events (participants affected / at risk) | 0/3517 | 0/37776

LIMITATIONS AND CAVEATS:
This study had the following limitations: 1) observational and therefore subject to unmeasured confounding; 2) utilized a claims based diagnosis of bipolar disorder (not gold standard); 3) not generalizable to low-income people with bipolar disorder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT02560701/Prot_SAP_000.pdf